CLINICAL TRIAL: NCT03120936
Title: The Stay Study: A Demonstration Project Advancing PrEP Delivery in the San Francisco Bay Area Transgender Community
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Public Health Foundation Enterprises, Inc. (Other)
Collaborators: San Francisco Department of Public Health (Other Government); University of California, San Francisco (Other); San Francisco Community Health Center (Unknown); Tri-City Health Center (Unknown); California HIV/AIDS Research Program (Other)
Responsible Party: Principal Investigator, Albert Liu, Clinical Research Director, Public Health Foundation Enterprises, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16-20339; PR15-SFDPH-026 (Other Grant/Funding Number: California HIV/AIDS Research Program)
Record Dates: First submitted 2017-04-11; First posted 2017-04-19 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Transgender Persons; Pre-Exposure Prophylaxis
Keywords: Adherence; Transgender; PrEP; HIV Prevention; Truvada; HIV Risk Reduction
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Main (Other): Emtricitabine / Tenofovir Disoproxil Oral Tablet and PrEP support.
  Interventions: Drug: Emtricitabine / Tenofovir Disoproxil Oral Tablet; Behavioral: PrEP support

INTERVENTIONS:
Drug: Emtricitabine / Tenofovir Disoproxil Oral Tablet — Open-label emtricitabine 200mg/tenofovir 300mg
  Other Names: Truvada; PrEP
Behavioral: PrEP support — HIV/STI testing and counseling, adherence counseling, medical exams, safety monitoring, short message system (SMS), ie text message, and peer support, panel management.

SUMMARY:
The Stay Study is a multi-site, open-label HIV pre-exposure prophylaxis (PrEP) demonstration project for advancing PrEP delivery in the San Francisco Bay Area Transgender Community. Approximately 188 HIV-uninfected participants will be enrolled at 4 sites in San Francisco and Fremont and will be provided Truvada to take orally once daily as PrEP.

DETAILED DESCRIPTION:
PrEP stands for Pre-Exposure Prophylaxis, an HIV prevention method that involves HIV negative people taking antiviral drugs daily to try to help prevent HIV infection. Studies with men who have sex with men (MSM) and transgender women showed that people who took PrEP were less likely to become infected with HIV than those who did not take it.

The main purpose of this PrEP Demonstration Project is to make PrEP accessible to people in the transgender community. As part of this project, we will study whether transgender women and men are interested in taking PrEP, and, if so, for how long and how frequently they take the medication and how these relate to demographics (such as race, age, and education). We will also assess reasons for stopping PrEP and measure sexual behaviors of participants in the demonstration project.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as a transgender woman, transgender man, or gender non-conforming
* Willing and able to provide written informed consent;
* Age ≥ 18 years;
* HIV-1-uninfected defined per site HIV testing algorithm performed within 7 (and up to 14) days of enrollment if PrEP naïve or within 90 days if currently on PrEP (see SSP manual)
* Expressed desired to use or continue PrEP, anticipated risk, or evidence of risk for acquiring HIV-1 infection including having any cisgender male or transgender female partners in the past 12 months and not in a mutually monogamous partnership with a recently tested, HIV-negative partner AND at least one of the following;

  1. any anal or vaginal sex in the past 12 months; or
  2. any STI diagnosed or reported in the past 12 months; or
  3. an ongoing sexual relationship with an HIV-positive partner; or
  4. exchange of money, gifts, shelter, or drugs for sex
* Fluent in English or Spanish

Exclusion Criteria:

* Individuals with any of the following will be excluded:

  * confirmed HIV infection by laboratory testing
  * clinical symptoms consistent with possible acute HIV infection [fatigue, fever, rash, night sweats, and adenopathy];
  * underlying bone disease (osteopenia or osteoporosis)
  * Receipt of prohibited medications: interleukin therapy, medications with significant nephrotoxic potential (including but not limited to amphotericin B, aminoglycosides, cidofovir, foscarnet and systemic chemotherapy), and medications that may inhibit or compete for elimination via active renal tubular secretion (including but not limited to probenecid)
  * No prior or current participation in the active arm of an HIV vaccine trial with evidence of vaccine-induced seropositivity.
  * Unwilling to attend quarterly follow-up visits, which will include risk reduction/adherence counseling and repeat laboratory testing
  * Has any other condition that, based on the opinion of the investigator or designee, would preclude provision of informed consent; make participation in the project unsafe; complicate interpretation of outcome data; or otherwise interfere with achieving the project objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender or gender non-conforming
Enrollment: 158 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
PrEP uptake and its correlates by gender identity, race/ethnicity, age, education, site, hormone status, and risk practices | Baseline
  Combined analysis of PrEP acceptance and refusal rates and sociodemographic correlates of PrEP acceptance and refusal.
Patterns and correlates of PrEP adherence among transgender individuals in the Stay Study. | 12 months
  Combined analysis of PrEP adherence rates as measured by: Tenofovir-diphosphate (TFV-DP) levels in dried blood spots (DBS); medication possession ratio; self-reported adherence. Patterns and correlates of adherence

SECONDARY OUTCOMES:
Reasons transgender people choose to initiate PrEP | Baseline
  Reasons for initiating PrEP
Reasons transgender people choose to decline PrEP | Baseline
  Reasons for declining PrEP
Measure of changes in sexual risk taking behavior among Stay Study participants taking PrEP | 12 months
  Computer-Assisted Self-interview (CASI) data: Numbers of sexual partners, by serostatus and condom use, and anal/vaginal sex episodes, by partner serostatus, role of respondent, and condom use; sexually transmitted infection (STI) testing
Measure of changes in STI among Stay Study participants taking PrEP | 12 months
  STI testing
Side effects and toxicities of PrEP among study participants | 12 months
  Combined analysis of side effects and toxicities, including creatinine elevations
PrEP discontinuations and reasons for discontinuation | 12 months
  PrEP discontinuations, reasons for discontinuation
Differences in duration of PrEP use and study retention by sociodemographics, including race/ethnicity, age, education and risk practices | 15 months
  Combined analysis of CASI and interview data.
The number of seroconversions and HIV drug resistance patterns among persons who become HIV infected in the project | 12 months
  HIV drug resistance patterns among persons who become infected
Effects of PrEP on hormone levels | 12 months
  Combined analysis of hormone levels as relates to measures of adherence, such as TFV-DP in DBS, tenofovir levels in plasma
The effect of hormone use on tenofovir-diphosphate concentrations among study participants | 12 months
  Combined analysis of hormone levels as relates to measures of adherence, such as TFV-DP in DBS, tenofovir levels in plasma
Social harms experienced by study participants | 12 months
  Social Impact questionnaire
Social benefits experienced by study participants | 12 months
  Social impact questionnaire
Referrals to other HIV prevention services within the Stay Study | 15 months
  Combined analysis of CASI and interview data
Access to and uptake of PrEP after project completion | 3 months
  Combined analysis of the proportion of participants interested in continuing PrEP and successfully able to access PrEP
Acceptability and uptake of Stay Study PrEP support components | 12 months
  Combined analysis of CASI and interview responses.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Y Liu, MD, MPH, Principal Investigator — Bridge HIV, San Francisco Department of Public Health; Erin Wilson, DrPH, Principal Investigator — Center for Public Health Research, San Francisco Department of Public Health
Locations (5):
- United States (5):
  - Tri-City Health Center, Fremont, California
  - Bridge HIV, San Francisco Department of Public Health, San Francisco, California
  - Tom Waddell Urban Health Clinic, San Francisco, California
  - San Francisco Community Health Clinic, San Francisco, California
  - Castro-Mission Health Center, San Francisco, California

IPD SHARING:
Plan to Share IPD: No